CLINICAL TRIAL: NCT01438125
Title: A Pilot Study to Evaluate the Safety and Preliminary Efficacy of MF-4181 for the Reduction of Scars Secondary to Abdominoplasty or Laparoscopy/Laparotomy Gynecologic Procedures
Brief Title: MF-4181 for the Reduction of Scars Secondary to Abdominoplasty or Laparoscopy/Laparotomy Gynecologic Procedures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Halscion, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAL-0082
Record Dates: First submitted 2011-09-20; First posted 2011-09-21 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Scars
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MF-4181 (Active Comparator): Scar halves randomized to treatment with device, opposite side treated per standard of care
  Interventions: Other: MF-4181
- Standard surgical wound closure (Active Comparator)
  Interventions: Other: Standard surgical wound closure

INTERVENTIONS:
Other: MF-4181 — Surgical procedure will be performed as per the standard of care. Scar halves randomized to treatment with device (MF-4181), opposite side treated per standard of care.
  Other Names: Hydrogel scaffold
  Arms: MF-4181
Other: Standard surgical wound closure — Surgical procedure will be performed as per the standard of care. Scar halves randomized to treatment with device (MF-4181), opposite side treated per standard of care.
  Arms: Standard surgical wound closure

SUMMARY:
The objective of the study is to evaluate the safety and preliminary efficacy of MF-4181, a hydrogel scaffold, in improving scars and their resulting consequences following abdominoplasty or laparoscopy/laparotomy gynecologic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 60 years of age undergoing abdominoplasty without intraoperative flexion at time of skin excision OR female subjects between 18 and 60 years of age undergoing diagnostic and/or operative laparoscopy/laparotomy gynecologic procedures.
* Weight between 50 and 95 kg with BMI between 20 and 30
* Able and willing to give written informed consent
* Willing to comply with the follow-up schedule

Exclusion Criteria:

* Need of concomitant surgical procedures that would be performed at the same time as the index surgical procedure or that would influence the healing process
* Previous abdominal surgery with scars or adhesions that would limit or complicate the index surgical procedure
* Presence of ventral or umbilical hernia requiring the use of prosthetic material
* Heart disease
* Pregnant or planning to become pregnant during the course of the study; the exception to this exclusion is if ectopic pregnancy is the reason for the procedure
* History of coagulopathy or bleeding disorder
* An American Society of Anesthesiologists (ASA) Score of >II
* Known diabetes
* Current or history of heavy smoking (i.e., 10 pack years)
* Active skin disorder or other condition that may interfere with healing or history of such a condition
* Planned use of an ON-Q® pain control device (I-Flow Corporation, Lake Forest, CA) or similar incisional intervention post index procedure
* Active collagen vascular disease or vasculitis, e.g., systemic lupus erythematosus, polyarteritis, dermatomyositis, systemic scleroderma or thrombotic thrombocytopenic purpura
* Anticipated use of DERMABOND® or another topical skin adhesive type of wound closure
* Unwilling or unable to return for follow-up visits
* Regular, continuous use of systemic corticosteroid therapy or topical corticosteroid use in the area to be treated
* Current participation or participation within the last 3 months in the study of an investigational drug, device, or biologic
* Unable or unwilling to follow post-operative instructions
* Known hypersensitivity to MF-4181, dextran, or any of its constituent materials
* Previous participation in this study to avoid multiple enrollments of an individual subject.
* Chemotherapy or hormone therapy for cancer within the last 3 months, or probability that these treatments will be required during the 6 months of study participation.
* Current or past radiation therapy in the abdominal incision

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Safety, defined as the absence of device related serious adverse events at 3 months post last MF-4181 treatment | 3 Months

SECONDARY OUTCOMES:
Investigator and Subject Observer Scar Assessment Scale (POSAS) | 12 months
Investigator and Subject Anchored Visual Analog Scar Evaluation Scale | 12 Months
Digital photographs evaluated by independent medical experts | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Wlodzimierz Baranowski, MD, Principal Investigator — Unaffliated
Locations (3):
- Poland (3):
  - II Katedra i Klinika Ginekologii Onkologicznej i Ginekologii, Lublin
  - Klinika Ginekologii Operacyjnej, Lublin
  - Klinika Ginekologii i Ginekologii Onkologicznej, Warsaw